CLINICAL TRIAL: NCT00758810
Title: Impact at One Year of a Secondary Prevention Educational Program on Cardiovascular Risk Factors, Daily Physical Activity, Dietary Habits and Blood Glucose and Fatty Acids in Coronary Syndromes Patients
Brief Title: Impact at One Year of a Secondary Prevention Educational Program on Cardiovascular Risk Factors
Acronym: OLIMPIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Alexis CERISIER, CHU de Saint-Etienne
Other Study IDs: 0608999
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome
Keywords: Health Education; Myocardial Infarction; Acute Coronary Syndrome; Quality of Life
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Health Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients without cardiac rehabilitation
- 2: Patients with cardiac rehabilitation

SUMMARY:
In secondary prevention, the beneficial role of cardiac rehabilitation programs after myocardial infarction, percutaneous coronary intervention or coronary artery bypass is now well established. The large majority of patients don't benefit from cardiac rehabilitation but for those who do, they usually follow an inhospital short health educational program with a sensibilisation to different coronary risk factors like smoking, overweight and inactivity. The impact of these inhospital short health educational programs combined to cardiac rehabilitation has never been totally evaluated, especially the impact on smoking cessation, weight loss and daily physical activity.

Therefore, the present study aims to evaluate the impact at one year on 400 consecutive patients' coronary risk profile of:

* an inhospital short health educational program alone
* an inhospital short health educational program combined to cardiac rehabilitation
* a cardiac rehabilitation program alone

DETAILED DESCRIPTION:
Classical CV risk factors, quality of life, daily physical activity and energy expenditure, smoking dependency and a daily quantification of fat intake are assessed with previously validated self-administrated questionnaires. Further factors like the lipid profile and glycaemia (with HbA1c in case of diabetes) will also be assessed. These evaluation will take place once at the of the hospitalization for acute coronary events in all patients, once at the end of any of the three rehabilitation programs for the concerned patients and, finally, one year after the hospitalization or the end of the rehabilitation program (mailed questionnaires and biological check-up). At this time, smoking dependency, medication, body mass index, any coronary event or need of coronary revascularization along with the professional ongoing situation (return to work) will be investigated.

As this study aims to evaluate the efficiency of France's clinical practice in spotting most relevant risk factors, the results of the present study could help us to focus the medical and paramedical resources on the modification of specific relevant risk factors.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome or myocardial infarcts

Exclusion Criteria:

* misunderstand the questionnaires
* living in institution
* severe morbidity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute coronary syndrome or myocardial infarctus
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2006-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
state of secondary prevention measures : Serum (fasting glucose, total cholesterol, HDL and LDL cholesterol, triglycerides, CPK, creatin), nutritional questionnaire, smoking cessation and physical activity | Inclusion and M12

CONTACTS AND LOCATIONS:
Overall Officials: Alexis CERISIER, MD, Principal Investigator — CHU de Saint-Etienne
Locations (4):
- France (4):
  - CH de Feurs, Feurs
  - CH de Firminy, Firminy
  - Centre Médical de Chavanne, Saint-Chamond
  - CHU de Saint-Etienne, Saint-Etienne

REFERENCES:
- [Background] De Backer G, Ambrosioni E, Borch-Johnsen K, Brotons C, Cifkova R, Dallongeville J, Ebrahim S, Faergeman O, Graham I, Mancia G, Manger Cats V, Orth-Gomer K, Perk J, Pyorala K, Rodicio JL, Sans S, Sansoy V, Sechtem U, Silber S, Thomsen T, Wood D; Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. European guidelines on cardiovascular disease prevention in clinical practice. Third Joint Task Force of European and Other Societies on Cardiovascular Disease Prevention in Clinical Practice. Eur Heart J. 2003 Sep;24(17):1601-10. doi: 10.1016/s0195-668x(03)00347-6. No abstract available. PMID 12964575
- [Background] AHA; ACC; National Heart, Lung, and Blood Institute; Smith SC Jr, Allen J, Blair SN, Bonow RO, Brass LM, Fonarow GC, Grundy SM, Hiratzka L, Jones D, Krumholz HM, Mosca L, Pearson T, Pfeffer MA, Taubert KA. AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update endorsed by the National Heart, Lung, and Blood Institute. J Am Coll Cardiol. 2006 May 16;47(10):2130-9. doi: 10.1016/j.jacc.2006.04.026. No abstract available. PMID 16697342
- [Background] Balady GJ, Williams MA, Ades PA, Bittner V, Comoss P, Foody JM, Franklin B, Sanderson B, Southard D; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; American Heart Association Council on Cardiovascular Nursing; American Heart Association Council on Epidemiology and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Association of Cardiovascular and Pulmonary Rehabilitation. Core components of cardiac rehabilitation/secondary prevention programs: 2007 update: a scientific statement from the American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee, the Council on Clinical Cardiology; the Councils on Cardiovascular Nursing, Epidemiology and Prevention, and Nutrition, Physical Activity, and Metabolism; and the American Association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2007 May 22;115(20):2675-82. doi: 10.1161/CIRCULATIONAHA.106.180945. Epub 2007 May 18. PMID 17513578